CLINICAL TRIAL: NCT04703361
Title: Effects of Ketones and Niacin in Heart Failure Patients
Acronym: KETO-COX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1010
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2020-10

CONDITIONS: Heart Failure, Systolic; Ketonemia
MeSH Terms: conditions — Heart Failure, Systolic; Ketosis | interventions — Niacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Niacin (Experimental): 12 patients with Heart failure with reduced ejection fraction (HFrEF) investigated with echocardiography and right heart catheterization.
  Interventions: Biological: Placebo NaCl; Biological: Niacin
- Na-3-OHB (Experimental): 12 patients with Heart failure with reduced ejection fraction (HFrEF) investigated with echocardiography and right heart catheterization.
  All patients will receive Aspirin before intervention and randomization.
  Interventions: Biological: Placebo NaCl; Biological: Na-3-OHB

INTERVENTIONS:
Biological: Placebo NaCl — Placebo
Biological: Niacin — B3 vitamin, Niacin
  Arms: Niacin
Biological: Na-3-OHB — Na-3-OHB
  Arms: Na-3-OHB

SUMMARY:
Ketones, 3-hydroxybutyrate (3-OHB), have shown to have beneficial hemodynamics effect in patients with hearth failure with reduced ejection fraction. The mechanisms behind these marked hemodynamic effects are currently unknown, but could involve prostaglandin-release. 3-OHB is the endogenous ligand for the G protein-coupled receptor hydroxy-carboxylic acid 2 (HCA2) receptor. This receptor has proven downstream effects on cAMP and systemic effects via release of prostaglandins.

In this present study we will investigate the cardiovascular effects of HCA2-receptor stimulation in heart failure patients.

DETAILED DESCRIPTION:
Heart Failure (HF) is a major public health issue because the disease affects 1-2% of the Western population and the lifetime risk of HF is 20%. HF is responsible for 1-2% of all healthcare expenditures and 5% of all hospital admissions. The cornerstone in the medical treatment of chronic HF is a combination of ACE-inhibitors/ATII-receptor antagonists, beta-blockers and mineralocorticoid receptor antagonists. Despite major improvements in the management and care of patients with HF, the 1-year mortality in patients with HF is 13 % 4 and >50% of HF-patients are admitted within a 2.5 year period 5. Furthermore, patients with HF have markedly decreased physical capacity and quality of life. Thus, there is a need for new treatment modalities in this group of patients.

Ketone bodies are produced in the liver and are crucial for energy generation during fasting in the heart and brain during, exercise and severe illnesses. However, ketosis can be safely obtained using dietary supplements and can increase exercise capacity in athletes. The most important ketone bodies are 3-hydroxybutyrate (3-OHB) and acetoacetate. Recently, it was demonstrated that patients with severe HF have increased myocardial utilization of the ketone body 3-OHB. It has been hypothesized that ketone bodies may act as a "superfuel" for the failing heart. In support of this, the glucose-lowering SGLT-2 inhibitor empagliflozin reduces the risk of hospitalizations and cardiovascular death in diabetic patients with HF and also increases circulating levels of 3-OHB.

By Positron Emission Tomography (PET) we have shown that ketone body infusion reduces myocardial glucose uptake and increases myocardial blood flow in healthy subjects. Data from another study conducted by our group show a 40% increase in cardiac output during infusion of 3-OHB. The mechanisms behind these marked hemodynamic effects are currently unknown, but could involve prostaglandin-release. 3-OHB is the endogenous ligand for the G protein-coupled receptor hydroxy-carboxylic acid 2 (HCA2) receptor. This receptor has proven downstream effects on cAMP and systemic effects via release of prostaglandins.

3-OHB have affinity to the HCA2 receptor and possibly a downstream effect resulting in the release of prostaglandins. The prostaglandin synthesis is dependent of cyclooxygenase (COX) enzyme, which can be inhibited by aspirin (ASA).

Niacin, vitamin B3, has been used as a treatment for dyslipidemia. Niacin is also a ligand for HCA2 receptor and the downstream release of prostaglandin cause side effects such as cutaneous flushing.

In this study we will investigate the cardiovascular effects of HCA2-receptor stimulation in heart failure patients. This will be done by comparing infusion of 3-OHB (preceded with ASA) and niacin.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure, Age ≥ 18 years old, LVEF ≤40%, New York Heart Association (NYHA) classification 2-3, Negative urine-HCG for women of childbearing potential, Ability to understand the written patient information and to give informed consent.

Exclusion Criteria:

* Symptomatic cardiac valve disease, Signs or history of major myocardial infarction (STEMI) within 1 month, Insulin treatment, Other disease or treatment making subject unsuitable for study participation as judged by the investigator.

Significant liver disease (defined by serum levels of alanine aminotransferase (ALAT) above 3 x upper limit of normal).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | 3 hours
  L/min

SECONDARY OUTCOMES:
Mixed venous saturation | 3 hours
  SvO2
Pulmonary wedge pressure | 3 hours
  PWR
Left ventricular ejection fraction | 3 hours
  EF
Circulating prostaglandin levels | 3 hours
  prostaglandins

CONTACTS AND LOCATIONS:
Overall Officials: Nigopan Gopalasingam, MD, Principal Investigator — University of Aarhus; Henrik Wiggers, MD, PhD, DMSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gopalasingam N, Christensen KH, Berg Hansen K, Nielsen R, Johannsen M, Gormsen LC, Boedtkjer E, Norregaard R, Moller N, Wiggers H. Stimulation of the Hydroxycarboxylic Acid Receptor 2 With the Ketone Body 3-Hydroxybutyrate and Niacin in Patients With Chronic Heart Failure: Hemodynamic and Metabolic Effects. J Am Heart Assoc. 2023 Jun 20;12(12):e029849. doi: 10.1161/JAHA.123.029849. Epub 2023 Jun 10. PMID 37301762